CLINICAL TRIAL: NCT05058495
Title: Investigation of the Effect of Mobile Lymphedema Self-Care Support Program on Self-Care, Quality of Life and Lymphedema-Related Symptoms in Women With Breast Cancer-related Lymphedema: A Randomized Controlled Trial
Brief Title: The Effect of Mobile Lymphedema Self-Care Support Program on Self-Care in Women With Breast Cancer-related Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Zeynep Deveci, Principal Investigator, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2020.KB.SAG.069
Record Dates: First submitted 2021-02-15; First posted 2021-09-27 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer Related Lymphedema
Keywords: self-care; mobile application; quality of life; patient education; symptoms; Breast Cancer Related Lymphedema
MeSH Terms: conditions — Breast Cancer Lymphedema

STUDY DESIGN:
Intervention Model Description: a prospective, randomized controlled study
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients were blinded and the person responsible for the data analysis will be masked as to the patient grouping for analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mobile programme users (Experimental): Patients will receive and use Mobile Lymphedema Self-Care Support Program application and will receive standart lymphedema education.
  Interventions: Other: Mobile Lymphedema Self-Care Support Program; Other: standart lymphedema education
- control group (Active Comparator): Patients who will receive standart lymphedema education
  Interventions: Other: standart lymphedema education

INTERVENTIONS:
Other: Mobile Lymphedema Self-Care Support Program — The Mobile Lymphedema Self-Care Support Program is composed of three section. First section includes the information about lymphedema and lymphedema self care. Second section includes the exercises videos which women can concurrently exercise with application and an alarm to remind to exercise. Last section is a social network form the women could chat and share anything with eachother. Patients will be told how to use the Mobile Lymphedema Self-Care Support Program and a contact number will be provided to ask questions about the program at any time.
  Other Names: standard lymphedema education
  Arms: mobile programme users
Other: standart lymphedema education — The control group will receive standard lymphedema education. The standard lymphedema education is an online education composed of information about lymphedema and lymphedema self-care.

SUMMARY:
The aim of this randomized controlled study is to evaluate the effect of the mobile lymphedema self-care support program on self-care, quality of life and symptoms related to lymphedema in women with breast cancer-related lymphedema.

H1: There is a difference between the Lymphedema Self-Care Scale mean score in women who develop lymphedema due to breast cancer, according to the use of the mobile lymphedema self-care support program.

H2: There is a difference between the Lymphedema Quality of Life Scale average score in women who develop lymphedema due to breast cancer according to the status of using the mobile lymphedema self-care support program.

H4: There is a difference between lymphedema arm circumference measurements according to the use of the mobile lymphedema self-care support program in women who develop lymphedema due to breast cancer.

H5: In women who develop lymphedema due to breast cancer, there is a difference in the situation of experiencing symptoms related to lymphedema according to the use of the mobile lymphedema self-care support program.

DETAILED DESCRIPTION:
The content of the mobile program was developed by the researchers. The mobile lymphedema self-care support program content was reviewed by an expert group consisting of doctors, physiotherapists and nurses working with patients with lymphedema. Patients will be contacted via telephone and will be informed about the study, and the experimental and control groups will be selected through the randomization program among the patients who agree to participate in the study and meet the sampling inclusion criteria. Patients were blinded, and blindness will be achieved in the data analysing stage. All measurements will be made to the experimental and control groups at the same time. The standard lymphedema self-care training will be given to the experimental and the control group. And the experimental group will be educated on how to use the mobile program. When the study is completed, the control group will also be allowed to use the mobile program.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as breast cancer-related lymphedema
* literate,
* having a smart phone,
* completed breast cancer treatment at least six months ago
* volunteering to participate in the study

Exclusion Criteria:

* having morbid obesity
* having metastazis
* having dementia
* having other psychiatric conditions
* another health problem that could prevent to exercise
* not using smart phone

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Breast Cancer Related Lymphedema Self-Care Scale Score | baseline, 1 month, 3 month
  The Breast Related Lymphedema Self-Care Scale is valid and reliable tool. The lowest score is 31, the highest score is 124. Higher scores indicate better self-care.
Change in Quality of Life Measure for Limb Lymphedema-Arm Scale Score | baseline, 1 month, 3 month
  The Quality of Life Measure for Limb Lymphedema-Arm Scale was translated and cross-culturally adapted to Turkish. The highest score of the scale is 80 and the lowest score is 20. A high score indicates poor quality of life.
Change in Lymphedema Symptom Intensity and Distress Survey Score | baseline, 1 month, 3 month
  The Turkish version of Lymphedema Symptom Intensity and Distress Survey is valid and reliable. The highest score of the scale is 30 and the lowest score is zero. A high score means experiencing too many symptoms.

SECONDARY OUTCOMES:
Change in Arm circumferences | baseline, 1 month, 3 month
  Circumferential measurements are taken at the metacarpal joint, wrist, elbow, 10 cm below and 10 cm above the elbow.

CONTACTS AND LOCATIONS:
Overall Officials: Özgül Karayurt, PhD, Study Chair — Izmir University of Economics; Sibel Eyigör, MD, Study Chair — Ege University
Locations (1):
- Ege Universitesi, Lymphedema unit of Physical therapy and rehabilitation department, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No